CLINICAL TRIAL: NCT03454568
Title: Measuring Cognition, Physical Function, and Quality of Life After Hematopoietic Cell Transplantation in Adults >/= 60 Years: A Feasibility Study
Brief Title: The Patients' Experience After Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0431-17-EP
Record Dates: First submitted 2018-01-19; First posted 2018-03-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Stem Cell Transplant Complications
Keywords: Stem Cell Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A saliva sample will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will examine how adults ≥ 60 years old thinking and memory abilities are affected by stem cell transplant; whether these changes affect day-to-day activities and quality of life and how thinking and memory abilities are affected by genetics, depression, anxiety and physical function. Genetics and other factors may affect the brain's chemicals or structure, and may increase risk for negative effects on thinking and memory.

DETAILED DESCRIPTION:
In this study, the investigators are looking to understand: 1) how adults ≥ 60 years old thinking and memory abilities are affected by stem cell transplant; 2) whether these changes affect day-to-day activities and quality of life; and 3) how thinking and memory abilities are affected by genetics, depression, anxiety and physical function. Genetics and other factors may affect the brain's chemicals or structure, and may increase risk for negative effects on thinking and memory. Participants will undergo neurocognitive testing along with the collection of a saliva sample and completing a battery of questionnaires and assessments.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 60-85
* Diagnosed with a hematological malignancy
* Is considering an autologous or allogeneic stem cell transplant OR has undergone stem cell transplant in the past 12 months and seen by the PI for pre-transplant evaluation.
* Is able to read, write, speak, and understand English

Exclusion Criteria:

* As per self report or medical record, history of central nervous system involvement and/or history of cranial irradiation or intrathecal chemotherapy except for patients with history of prophylactic intrathecal chemotherapy.
* As per self report or medical record, history of stroke, head injury, neurosurgery, seizure disorder, or demyelinating disorder.
* As per self report or medical record, history of substance use disorder.
* As per self report or in the judgement of the consenting professional, uncorrected vision loss.
* As per self report or medical record, primary psychiatric disorder necessitating inpatient treatment in the last 12 months.
* As per self report or medical record, history of allogeneic and or autologous stem cell transplant.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is being recruited from the Fred & Pamela Buffett Cancer Center at the University of Nebraska Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Assess differences with cognitive function in older patients undergoing allogeneic or autologous stem cell transplant at 4 timepoints. | Before transplant; Post Transplant at 100 days, 6 months, and 12 months
  Cognition will be measured using a neuropsychological battery.

SECONDARY OUTCOMES:
Assess quality of life of of older patients undergoing allogeneic and autologous transplant at 4 timepoints. | Before transplant; Post Transplant at 100 days, 6 months, and 12 months
  Quality of life will be measured with the EORTC Quality of Life-30C questionnaire.
Assess activity engagement of older patients undergoing allogeneic and autologous transplant at 4 timepoints. | Before transplant; Post Transplant at 100 days, 6 months, and 12 months
  Activity engagement will be measured with the Activity Card Sort-modified.
Describe genetic variations in genes potentially involved in cognitive function and cancer treatment. | 1 time collection: Before transplant
  A saliva sample will be collected to look at genetic variations.

CONTACTS AND LOCATIONS:
Overall Officials: Thuy Koll, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03454568/ICF_000.pdf